CLINICAL TRIAL: NCT02464007
Title: A Phase 1 Study of rSIFN-co for Subjects With Advanced Solid Tumors Where Interferons Are Known to Have Demonstrated Antitumor Activity
Brief Title: Study of rSIFN-co for Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol has been amended and the Protocol amendment of Phase II was approved by the US FDA on Nov 2024 through SN0028.
Sponsor: Sichuan Huiyang Life Science and Technology Corporation (Industry)
Collaborators: Medelis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STM-04
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2024-04

CONDITIONS: Malignancies Including Melanoma, Kidney, Lung, Colorectal, Prostate, Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sSIFN-co (Experimental): Dose escalation of rSIFN-co
  Interventions: Biological: rSIFN-co

INTERVENTIONS:
Biological: rSIFN-co — Artificial recombinant super-compound interferon (rSIFN-co) is a product of patented technological research made possible through protein modulation by spatial conformation control technology, and was developed by Sichuan Huiyang Life Science and Technology Corporation.

SUMMARY:
In this EffTox dose escalation study, up to 3 dose levels will be tested. The optimal dose (OD) of rSIFN-co will be determined using the EffTox design. Additional subject cohorts will not be enrolled until all subjects at the current dose level complete 28 days without DLT. The optimal dose (OD) will be determined by evaluation of safety in each cohort and disease response by RECIST 1.1 at 8 weeks. Once the OD is determined, enrollment will continue until at least 9 subjects total are accrued at the OD. Pharmacokinetics of rSIFN-co will be conducted for all tested dose levels to characterize dose proportionality.

DETAILED DESCRIPTION:
The initial cohort will be 3 subjects. Escalation to the next dose will continue unless a subject experiences a DLT, at which time a cohort will be expanded to up to 6 subjects. Provided there is only one DLT in that cohort, the dose will be escalated. However, if there are 2 DLTs in that cohort of up to 6 subjects, previous dose level will be expanded to total of 9 subjects.

If none of the dose levels are acceptable at study completion (i.e., >33% of subjects experiencing a DLT), an OD will not be identified, and the drug does not warrant further investigation.

ELIGIBILITY:
Inclusion Criteria

1. Male or female ≥ 18 years of age
2. Diagnosis of advanced solid tumors limited to: melanoma, kidney cancer, lung cancer, colorectal carcinoma, prostate cancer, and neuroendocrine tumor progressing on standard therapy.
3. Has measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1.
4. Prior systemic chemotherapy, immunotherapy (including interferon), or biological therapy, radiation therapy and/or surgery for resection of solid tumor (limited to: melanoma, kidney cancer, lung cancer, colorectal carcinoma, prostate cancer, and neuroendocrine tumor) are allowed.
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
6. Has adequate hepatic function defined as total bilirubin ≤1.5 mg/dL, unless associated with hepatobiliary metastases or Gilbert syndrome, then total bilirubin or ≤ 2 ULN. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 x ULN for subjects with known hepatic metastases.
7. Has adequate renal function defined as serum creatinine or ≤ 1.5 × ULN and creatinine clearance or ≥ 40 ml/min.
8. Has adequate bone marrow function defined as a hemoglobin > 9 g/dL, absolute neutrophil count (ANC) ≥1.5 ×10⁹/L , and platelet count ≥100,000/mm³. For subjects who received chemotherapy for melanoma just prior to screening for the study subject needs to have a hemoglobin > 9 g/dL, absolute neutrophil count (ANC) >2 × 10⁹/L, and platelet count ≥100,000/mm³.
9. Must be willing and able to comply with study visits and procedures.
10. Has read, understood and signed the informed consent form (ICF) approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).
11. Women of childbearing potential (WOCP) must not be pregnant (confirmed by a negative pregnancy test, with a serum beta-HCG with a sensitivity of 50 mIU/ml within 7 days of study treatment) or breast-feeding. In addition, a medically acceptable method of birth control must be used such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence during the study and at least one month after the last dose of study drug. Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP.
12. Men who are not surgically or medically sterile must agree to use an acceptable method of contraception. Male subjects with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms from the date of the first dose of study drug through at least one month after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative.

Exclusion Criteria

1. Chemotherapy, immunotherapy (including interferon), or biological therapy, radiation therapy and/or surgery within 4 weeks prior to first dose of study drug.
2. Prior mTOR inhibitor therapy within 4 weeks prior to first dose of study drug.
3. Has a history of autoimmune disorders, including uncontrolled diabetes ("uncontrolled" defined as Hemoglobin A1c ≥ 9% in 28 days prior to study).
4. Chronic use of steroid therapy.
5. Has a history of epilepsy, depression or other psychiatric disorders.
6. Has a history of an arterial thromboembolic event within the prior six months including cerebrovascular accident, transient ischemic attack, myocardial infarction, or unstable angina.
7. Has uncontrolled human immunodeficiency virus (HIV) (defined as HIV RNA >500 copies/ml and CD4+ count<200/mm³ on antiretroviral therapy)infection, or hepatitis B (defined as ALT > 1 x ULN, and HBV DNA >2000 IU/ml), or hepatitis C (defined as ALT > 1 x ULN, persistent viremia on antiviral therapy) infections.
8. Has a history of blood clots, pulmonary embolism, or deep vein thrombosis unless controlled by anticoagulant treatment (patient must be on stable dose for 2 weeks).
9. Prior allogeneic bone marrow or organ transplantation.
10. Has any clinically significant infection, i.e., any acute viral, bacterial, or fungal infection that requires specific treatment (anti-infective treatment has to be completed ≥ 7 days prior to study entry).
11. Has any other severe, uncontrolled medical condition, including unstable congestive heart failure (Stage III-IV of the New York Heart Association Functional Classification) or has a known or suspected allergy to the study drug or any study drug component.
12. Pregnant or breastfeeding - interferon products (e.g., Infergen®) is Pregnancy Category C, (i.e., animal reproduction studies have shown an adverse effect on the fetus and there are no adequate and well-controlled studies in humans.). Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (β-HCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
13. Subject has received other investigational drugs within 14 days prior to first dose of study drug.
14. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for enrollment in this study.
15. Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinically significant or baseline prolongation of the rate-corrected QT interval (e.g., repeated demonstration of QTc interval > 480 milliseconds).
16. Presence of any non-healing wound, fracture, or ulcer within 28 days prior to the first dose of study drug.
17. Has any condition that, in the opinion of the investigator, might jeopardize the safety of the subject or interfere with protocol compliance.
18. Has any mental or medical condition that prevents the subject from giving informed consent or participating in the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2024-11 (Actual); Study Completion 2024-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28-days

CONTACTS AND LOCATIONS:
Overall Officials: Guangwen Wei, Study Director — Superlab
Locations (4):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Chicago, Illinois
  - HealthPartners Institute, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided
This has not been determined.